CLINICAL TRIAL: NCT06565676
Title: Effect of Whey Powder Added Bread on Postprandial Blood Glucose
Brief Title: Effect of Whey Powder Bread on Blood Glucose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Aslı Onur Canaydın, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: ERU-BD-AOC-01
Record Dates: First submitted 2024-08-08; First posted 2024-08-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Diet, Healthy
Keywords: Whey protein; Blood glucose; Enriched food; Sustainable nutrition
MeSH Terms: interventions — Bread

STUDY DESIGN:
Intervention Model Description: All volunteer participants were randomly assigned to a breakfast meal containing all types of bread (white flour bread, white flour bread with whey powder added, whole wheat flour bread and whole wheat flour bread with whey powder added) for four days.
Who Masked: Participant, Investigator
Masking Description: The order of bread types to be consumed by the participants will be determined by a person who is not a researcher in the study by simple randomization method using Microsoft Excel program. A researcher who does not interact with the participants will provide the participants with breakfast containing the test breads every day. Due to the difference in bread types, the comparison of breads will be double-blind. An investigator who does not know the type of bread consumed will be assigned for glucose measurement and will be blinded to the assigned bread.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- White Bread (Experimental): Participants will have their fasting blood glucose measured immediately before the meal containing the white flour test bread and will then be asked to consume the entire test bread with their breakfast meal within 15 minutes.
  Interventions: Dietary Supplement: Bread with whey protein powder added
- White Bread with Whey Powder (Experimental): Participants will have their fasting blood glucose measured immediately before the meal containing the white flour with added whey powder test bread and will then be asked to consume the entire test bread with their breakfast meal within 15 minutes.
  Interventions: Dietary Supplement: Bread with whey protein powder added
- Wheat Bread (Experimental): Participants will have their fasting blood glucose measured immediately before the meal containing the wheat flour test bread will then be asked to consume the entire test bread with their breakfast meal within 15 minutes.
  Interventions: Dietary Supplement: Bread with whey protein powder added
- Wheat Bread with Whey Powder (Experimental): Participants will have their fasting blood glucose measured immediately before the meal containing the wheat flour with added whey powder test bread and will then be asked to consume the entire test bread with their breakfast meal within 15 minutes.
  Interventions: Dietary Supplement: Bread with whey protein powder added

INTERVENTIONS:
Dietary Supplement: Bread with whey protein powder added — Volunteer participants will consume bread with and without whey powder added and its effect on blood sugar will be examined.

SUMMARY:
The aim of the study was to add whey powder, which is lost as waste in cheese production and has many health benefits, to bread, which is consumed very much daily in Turkey, to enrich bread in terms of nutrients and to examine the effect of whey powder added bread on postprandial blood glucose. In the study, all volunteer participants will be randomly assigned to a breakfast meal containing all types of bread (white flour bread, white flour bread with whey powder added, whole wheat flour bread and whole wheat flour bread with whey powder added) for four consecutive days and their blood glucose levels will be measured at certain minutes. There are no studies in the literature investigating the effect of whey powder added to bread on blood glucose.

DETAILED DESCRIPTION:
In cheese making, whey is the liquid that is separated from the clot formed as a result of coagulation of milk with rennet or acid, does not coagulate and contains milk dry matter. Serum proteins in whey increase the nutritional value of whey proteins and help the absorption of minerals. In addition to their nutritional value, whey proteins have important health effects in terms of other metabolic functions such as strengthening immunity, stimulating gastrointestinal hormone secretion, antiviral activity, and satiety response. Therefore, the aim of this study was to add whey powder, which is lost as waste in cheese production and has many health benefits, to bread, which is consumed very much daily in Turkey, to enrich bread in terms of nutrients and to examine the effect of whey powder added bread on postprandial blood glucose. The study is planned to be conducted in 20 healthy individuals aged 19-35 years with normal body mass index (18.5-25.0 kg/m2) between August 2024 and March 2025. In the study, all volunteer participants will be randomly assigned to a breakfast meal consisting of all bread types (bread made from white flour, bread made from white flour with whey powder added, bread made from whole wheat flour and bread made from whole wheat flour with whey powder added) for four consecutive days. During these days, participants will have their fasting blood glucose measured immediately before the meal containing the test bread and will then be asked to consume the entire test bread with their breakfast meal within 15 minutes. After breakfast, postprandial blood glucose will be measured at 15, 30, 45, 60, 90, 120 minutes. Food consumption records will be taken by the researchers and participants will be instructed not to eat or drink anything 8 hours before breakfast and not to perform any physical activity other than their daily activities during that day. Anthropometric measurements will be taken by the researchers using appropriate methods and food consumption records will be questioned in detail on a daily basis. According to the food consumption record, the types and amounts of foods consumed daily will be determined and energy, macro and micronutrient values will be analyzed using the Turkey Specific Nutrition Information System (BeBIS) computer program. There is no study in the literature investigating the effect of whey powder added to bread on blood glucose. In addition, enriching bread, which is very important in the nutrition of the Turkish nation, with whey powder, which is considered as "waste", will contribute to both sustainability and economy.

ELIGIBILITY:
Inclusion Criteria:

* having a normal BMI (18.5-25.0 kg/m2),
* being between 19-35 years of age,
* not having any chronic disease,
* not taking any medication, multivitamin or mineral supplements,
* not drinking alcohol or smoking,
* not engaging in heavy physical activity,
* not being pregnant or lactating.

Exclusion Criteria:

* having very low and high BMI (<18.5 kg/m2 and >25.0 kg/m2),
* being younger than 19 years and older than 35 years,
* having any chronic disease,
* taking medication, multivitamin or mineral supplements,
* alcohol and smoking, heavy physical activity,
* being pregnant or lactating

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose response | Two hours postprandial period (from fasting to 120 minutes after the test breakfast)
  Postprandial glucose response was quantified as incremental area under the curve (iAUC), which was calculated according to the trapezoidal rule by using serum glucose values at time points 0, 15, 30, 45, 60, 90, and 120 minutes. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı ONUR CANAYDIN, MsC, Principal Investigator — Erciyes Üniversitesi
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No